CLINICAL TRIAL: NCT01160666
Title: A Phase 2, Proof of Concept, 52-Week Open Study to Evaluate the Efficacy and Safety of Belimumab (HGS1006, LymphoStat-B™), a Fully Human Monoclonal Anti-BLyS (BAFF) Antibody, in Subjects With Primary Sjögren's Syndrome
Brief Title: Efficacy and Safety of Belimumab in Subjects With Primary Sjögren's Syndrome
Acronym: BELISS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Human Genome Sciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P090208
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-07

CONDITIONS: Sjögren's Syndrome
Keywords: Belimumab; Sjögren's syndrome; Sjögren disease
MeSH Terms: conditions — Sjogren's Syndrome | interventions — belimumab; Antibodies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1: Belilumab (Experimental)
  Interventions: Drug: Belimumab

INTERVENTIONS:
Drug: Belimumab — Belimumab will be administered at 10 mg/kg at Days 0, 14, 28 and then every 28 days until week 24 for all patients and week 48 for those considered responders at week 28.
  Other Names: HGS1006, LymphoStat-B™,; Human Monoclonal Anti-BLyS (BAFF) Antibody; Benlysta

SUMMARY:
Sjögren's syndrome (SS) is a systemic autoimmune disease characterized by an increase in BAFF (BLyS) levels and a resulting B cell hyperactivity. B cells are involved in the pathogenesis of SS in both systemic and glandular features, and B cell downregulation may lead to a decrease of disease activity. Moreover, pathogenesis of SS is closed to that of Systemic lupus erythematosus, where Belimumab has been proven to be effective.

DETAILED DESCRIPTION:
Sjögren's syndrome (SS) is a systemic autoimmune disease characterized by an increase in BAFF (BLyS) levels and a resulting B cell hyperactivity. B cells are involved in the pathogenesis of SS in both systemic and glandular features, and B cell downregulation may lead to a decrease of disease activity. Moreover, pathogenesis of SS is closed to that of Systemic lupus erythematosus, where Belimumab has been proven to be effective.

This phase II open-label study has 2 mains objectives:

* To evaluate the proof of concept of efficacy of belimumab in subjects with SS
* To evaluate the safety and tolerability of belimumab in subjects with SS Belimumab will be administered (10mg/kg on D0 D14 D28 and every 28 days for 24 weeks, with extension to 48 weeks if responders) to all patients

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of primary SS according to the updated American European Consensus Group Criteria. In addition, patients must be always positive for anti-SSA or anti-SSB antibodies
* Have the presence, at screening, of Systemic involvement (polysynovitis, skin, renal, lung, CNS involvement, peripheral neuropathy, vasculitis, autoimmune cytopenia, defined in Annex 1) or persistent (up to 2 months) parotid, submandibular or lachrymal gland swelling of more than 2 cm OR

Objective sicca (positive oral and/or ocular tests reported in the American European Consensus Group Criteria) with at least one among the following biological features of serum B lymphocyte activation :

increased IgG levels increased free light chain levels of immunoglobulins (according to central laboratory ranges) increased serum beta2-microglobulin levels decreased C4 levels (C4 levels inferior to central laboratory ranges) monoclonal gammapathy cryoglobulinemia OR

* SS of more recent onset, i.e., less than 5 years of duration of symptoms, associated with:

  * oral or ocular dryness
  * fatigue
  * musculoskeletal pain (i.e, 3 criteria for response as reported at page (ix-x), characterized by VAS score more than 50/100 in all the 3 fields.

Exclusion Criteria:

1. Any BLyS-targeted (BLyS-receptor fusion protein [BR3], TACI Fc, or belimumab) at any time.
2. Any of the following within 364 days of Day 0:

   * B-cell targeted therapy (eg, rituximab, other anti-CD20 agents, anti-CD22 [epratuzumab], anti-CD52 [alemtuzumab]
   * A biologic investigational agent other than B cell targeted therapy (eg, abetimus sodium, anti CD40L antibody [BG9588/ IDEC 131]).

4- Intravenous or oral cyclophosphamide within 180 days of Day 0.

5- Any of the following within 90 days of Day 0:

* Anti-TNF therapy
* Interleukin-1 receptor antagonist
* Abatacept
* Interleukin-6 receptor antagonist
* Intravenous immunoglobulin
* Prednisone > 100 mg/day
* Plasmapheresis.

  9- Very severe SS disease.

  10- Major organ or hematopoietic stem cell/marrow transplant.

  11- Unstable or uncontrolled acute or chronic diseases not due to SS

  13- History of malignant neoplasm within the last 5 years, except for adequately treated cancers of the skin (basal or squamous cell) or carcinoma in situ of the uterine cervix.

  14- Required management of acute or chronic infections, as follows:
* Currently on any suppressive therapy for a chronic infection
* Hospitalization for treatment of infection within 60 days of Day 0.
* Use of parenteral (IV or IM) antibiotics

  16- Historically or at screening positive test for HIV antibody, hepatitis C virus antibodies, or, hepatitis B surface antigen (HbsAg) (with or without positive serum HBV DNA), or antiHBcAg positivity (without anti-HbsAg positivity).

  17- Grade 3 or greater laboratory abnormality based on the protocol toxicity scale except for the following that are allowed:
* Stable Grade 3 prothrombin time (PT) secondary to warfarin treatment.
* Stable Grade 3/4 proteinuria (≤ 6 g/24 hour equivalent by spot urine protein to creatinine ratio allowed). (mentioned earlier in Exclusion #8)
* Stable Grade 3 neutropenia or stable Grade 3 white blood cell count.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
response rate | week 28
  A response is defined as the fulfilment of any 2 of the 5 following response criteria(values are compared to that of baseline [Day0]):
  * ≥ 30% reduction of the patient's dryness VAS
  * ≥ 30% reduction of the patient's fatigue VAS
  * ≥ 30% reduction of the patient's musculoskeletal pain VAS
  * ≥ 30% reduction of the physician's systemic activity VAS
  * ≥ 25% reduction of serum levels of any of the following B cell activation biomarkers (free light chains of immunoglobulin, beta2-microglobulin, monoclonal component, cryoglobulinemia, IgG) or ≥ 25% C4 increase

SECONDARY OUTCOMES:
safety and tolerability of belimumab | 52 weeks
  Evaluate the safety and tolerability of belimumab in subjects with SS

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Mariette, PhD, Principal Investigator — Rheumatology Department of BICETRE Hospital
Locations (1):
- Assistance Publique - Hôpitaux de Paris : BICETRE Hospital, Le Kremlin-Bicêtre, France

REFERENCES:
- [Derived] Bowman SJ, Fisher BA. Stratifying primary Sjogren's syndrome: killers in the balance? Arthritis Res Ther. 2015 Dec 7;17:351. doi: 10.1186/s13075-015-0878-9. PMID 26639390
- [Derived] Seror R, Nocturne G, Lazure T, Hendel-Chavez H, Desmoulins F, Belkhir R, Ravaud P, Benbijja M, Poirier-Colame V, Taoufik Y, Mariette X. Low numbers of blood and salivary natural killer cells are associated with a better response to belimumab in primary Sjogren's syndrome: results of the BELISS study. Arthritis Res Ther. 2015 Sep 4;17(1):241. doi: 10.1186/s13075-015-0750-y. PMID 26336930